CLINICAL TRIAL: NCT05085860
Title: Feasibility of Examining Acute Responses to Exercise in Symptomatic Females and Males With Atrial Fibrillation: a Pilot Randomized Crossover Study
Brief Title: Acute Responses to Exercise in Females and Males With Symptomatic Atrial Fibrillation
Acronym: ACUTE-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20210524-01H
Record Dates: First submitted 2021-09-13; First posted 2021-10-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Persistent Atrial Fibrillation; Paroxysmal Atrial Fibrillation
Keywords: Exercise; Sex differences; Pilot; Symptoms
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This is a repeated measures randomized counter-balanced design. All participants will complete three conditions in a randomized order, with a wash-out week in between.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate Intensity Continuous Training (MICT) (Experimental): Participants will do 3 sessions of moderate-intensity continous exercise training over 7 days
  Interventions: Behavioral: Moderate-intensity continuous training (MICT)
- High Intensity Interval Training (HIIT) (Experimental): Participants will do 3 sessions of high-intensity interval training over 7 days
  Interventions: Behavioral: High-intensity interval training (HIIT)
- Rest (No Intervention): Participants will abstain from doing moderate- to high-intensity interval training over 7 days

INTERVENTIONS:
Behavioral: Moderate-intensity continuous training (MICT) — Participants will engage in exercise and record AF symptoms prospectively over 7 days
  Arms: Moderate Intensity Continuous Training (MICT)
Behavioral: High-intensity interval training (HIIT) — Participants will engage in exercise and record AF symptoms prospectively over 7 days
  Arms: High Intensity Interval Training (HIIT)

SUMMARY:
The main purpose of this pilot project is to measure the feasibility of conducting a randomized crossover study examining short-term changes in atrial fibrillation (AF) symptoms in symptomatic females and males with paroxysmal or persistent AF when they engage in a standard week of exercise (i.e. moderate-intensity continuous training [MICT] or high-intensity interval training [HIIT]) compared to a control week (i.e. no moderate to vigorous exercise over 7 days).

DETAILED DESCRIPTION:
Exercise training (e.g. 8 to 12-week exercise programs) has been shown to improve cardiorespiratory fitness and QoL, and reduce atrial fibrillation (AF) symptoms and time in AF in patients with AF. However, regular exercise participation is hindered by patient concerns regarding an increase in AF symptoms and episodes during or following an exercise session. Patients with AF also worry about potential negative consequences of increasing heart rate during exercise. This fear may be sex-specific as females report more AF symptoms at rest, experience faster heart rates during exercise and AF, and report greater symptoms of fear/anxiety than males. How exercise acutely changes AF symptoms remains to be examined.

The main purpose of this pilot project is to measure the feasibility of conducting a randomized crossover study examining short-term changes in AF symptoms in symptomatic females and males with paroxysmal or persistent AF when they engage in a standard week of exercise (i.e. moderate-intensity continuous training [MICT] or high-intensity interval training [HIIT]) compared to a control week (i.e. no moderate to vigorous exercise over 7 days). As secondary outcomes we will explore sex differences in short-term changes in AF symptoms (self reported with a questionnaire) and AF status (device measured with a wireless four-finger AliveCor KardiaMobile ECG) when symptomatic patients with AF engage in a standard week of exercise (i.e. HIIT, MICT) compared to a control week. Results from this pilot study will provide novel insight into the typical acute response to exercise in females and males with AF, and will inform appropriate approaches for the conduct of a future larger trial. This work is key to informing practitioners and patients of the typical acute exercise response in the AF population with the goal of facilitating exercise prescription and participation.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal and Persistent AF
* Rate controlled (resting ventricular rate <110 bpm)
* Able to do a symptom limited exercise test
* At least 40 years of age
* Self-reports being symptomatic in the past 4 weeks
* If female, self-reports being post-menopausal
* Able to read and understand English or French
* Agrees to sign informed consent

Exclusion Criteria:

* Currently participating in routine exercise training
* Unstable angina or uncontrolled diabetes mellitus; or established diagnosis of severe mitral or aortic stenosis, or hypertrophic obstructive cardiomyopathy with significant obstruction
* Unable to access the Internet or a phone (iPhone and iPad require iOS version 10.0 and up, Android requires version 6.0 and up) during the study period
* Has an automated external defibrillator, an implantable cardioverter defibrillator or other types of pacemaker
* Unwilling or unable to complete the three conditions
* Unable to provide written, informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the pilot study - Recruitment and consent rate | Through study completion, an average of 1.5 years
Feasibility of the pilot study - Participant fidelity | During the week of HIIT and MICT (2 weeks)
  E.g. ability of participants to comply with the exercise prescription, number of exercise sessions attended
Feasibility of the pilot study - Study retention | Through study completion, an average of 1.5 years
  Dropout rate of participants
Feasibility of the pilot study - Study eligibility refinement | Through study completion, an average of 1.5 years
  Data to refine inclusion and exclusion criteria for a larger trial will be used by balancing safety, ability to complete the intervention, and generalizability (e.g. is an exclusion criterion of threshold of participation in >2 structured exercise sessions/week sufficient or restrictive?)
Feasibility of the pilot study - Adverse events | Through study completion, an average of 1.5 years
  Side effects and adverse events during the study

SECONDARY OUTCOMES:
AF symptoms self-reported with a 7-day patient symptom questionnaire | 3 weeks (1 week of HIIT, 1 week of MICT, 1 week fo rest)
  Secondary objectives will explore sex differences in short-term changes in AF symptoms when symptomatic females and males with AF engage in a standard week of exercise (MICT or HIIT), compared to a control (rest) week.
  Participants will report AF symptoms prospectively during each condition. They will complete a 7-day questionnaire during MICT, a 7-day questionnaire during HIIT and a 7-day questionnaire during the rest week.
AF status measured daily with a KardiaMobile device | 3 weeks (1 week of HIIT, 1 week of MICT, 1 week fo rest)
  Secondary objectives will explore sex differences in short-term changes in AF status when symptomatic females and males with AF engage in a standard week of exercise (MICT or HIIT), compared to a control week.
  AF status will be measured with a Kardiamobile AliveCor wireless device. Participants will be asked to record 3 x 30-second ECGs a day (morning, afternoon, evening) during each condition (MICT, HIIT and rest). The ECG recording will allow the identification of whether the participant is in sinus rhythm or in atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada